CLINICAL TRIAL: NCT05589714
Title: Universal Rare Gene Study: A Registry and Natural History Study of Retinal Dystrophies Associated With Rare Disease-Causing Genetic Variants
Acronym: Uni-Rare
Status: Recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: Uni-Rare
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: Inherited Retinal Degeneration; Retinitis Pigmentosa
Keywords: Inherited Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Younger Age Cohort: Participants ages ≥ 4 years and < 8 years old will be designated as the Younger Age Cohort.
  * Participants in this cohort will not be assigned a Vision Cohort.
  * Registry/Screening Visit and Natural History Study Visits will have an abbreviated testing schedule, detailed in the Schedule of Study Visits and Procedures table.
- Vision Cohort 1: Participants who are aged ≥ 8 years old will be designated into a Vision Cohort based on data in the better eye, at the Registry/Screening Visit. Criteria that must be met in the better eye* at the Registry/Screening Visit: visual acuity ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) and visual field** diameter 10 degrees or more in every meridian of the central field
- Vision Cohort 2: Participants who are aged ≥ 8 years old will be designated into a Vision Cohort based on data in the better eye, at the Registry/Screening Visit. Criteria that must be met in the better eye* at the Registry/Screening Visit: visual acuity ETDRS letter score of 19-53 (approximate Snellen equivalent 20/100 to 20/400) or visual acuity ETDRS letter score of 54 or more (approximate Snellen equivalent 20/80 or better) and visual field** diameter less than 10 degrees in any meridian of the central field
- Vision Cohort 3: Participants who are aged ≥ 8 years old will be designated into a Vision Cohort based on data in the better eye, at the Registry/Screening Visit. Criteria that must be met in the better eye* at the Registry/Screening Visit: visual acuity ETDRS letter score of 18 or less (approximate Snellen equivalent 20/500 or worse)

SUMMARY:
This is an international, multicenter study with two components:

Registry

* A standardized genetic screening and a prospective, standardized, cross-sectional clinical data collection
* Enrollment is open to all genes on the RD Rare Gene List

Natural History Study

* A prospective, standardized, longitudinal Natural History Study
* Enrollment opens gene-by-gene, based on funding and within-gene Registry enrollment The study objectives are as follows.

Registry Objectives

1. Genotype Characterization
2. Cross-Sectional Phenotype Characterization (within gene)
3. Establish a Link to My Retina Tracker Registry (MRTR)
4. Ancillary Exploratory Studies - Pooling of Genes

Natural History Study Objectives

1. Natural History (within gene)
2. Structure-Function Relationship (within gene)
3. Risk Factors for Progression (within gene)
4. Ancillary Exploratory Studies - Pooling of Genes

DETAILED DESCRIPTION:
This study includes multiple phases.

1. Screening Phase

   The patient's current genetic report will be reviewed. Genetic testing will not be performed in this study. A prior conclusive genetic test will be assessed for screening analysis. Having at least one gene on the RD Rare Gene List meets one of the eligible Genetic Screening Criteria and other eligibility criteria can be evaluated based on medical history.
2. Genetic Screening Phase:

   Genetic reports for participants enrolled into the genetic screening phase will be uploaded to study website for review and confirmation by Central Genetics Auditor (CGA) as meeting Genetic Screening Criteria.Participants confirmed as meeting those criteria will be considered enrolled into the Registry.
3. Registry Phase:

   The flow of participants who are enrolled into the Registry depends on whether their causal gene is designated as a Natural History Study (NHS) Target Gene. If they are not Designated as NHS Target Gene, they will receive annual phone calls up to 48 months from the Registry/Screening visit or until the gene is designated as NHS Target Gene. If they are Designated as NHS Target Gene participants will be considered pending enrollment into the NHS.

   The Registry will establish genetically and clinically well-characterized cohorts of patients across hundreds of genetic variants associated with retinal dystrophy (RD). Characterization of these patients will accelerate eligibility screening for the Natural History Study, provide cross-sectional data on phenotype-genotype associations, and contribute to our knowledge of pathogenicity of these rare disease-causing variants.
4. Natural History Study (NHS) Phase

Participants pending enrollment will return to the clinic for the NHS Enrollment/Baseline Visit and return to the clinic for follow-up visits.

The Natural History Study will accelerate the identification and development of sensitive, reliable outcome measures for clinical trials, which will facilitate development of treatments for retinal dystrophies due to disease-causing genetic variants. The expected impact of the Natural History Study is as follows:

1. Describe the natural history of retinal degeneration in patients with rare disease-causing genetic variants
2. Identify sensitive structural and functional outcome
3. Identify well-defined subpopulations for future clinical trials of investigative treatments for rare inherited retinal degeneration

ELIGIBILITY:
Inclusion Criteria: Participants must meet all the following inclusion criteria at the Registry/Screening Visit to be eligible to enroll into the genetic screening phase:

1. Willing to participate in the study and able to communicate consent during the consent process
2. Willing and able to complete all applicable Registry/Screening Visit assessments
3. Age ≥ 4 years
4. Must have a single gene on the RD Rare Gene List which meets one of the Genetic Screening Criteria below based on a genetic report* from a clinically certified lab (or from a research lab which has been approved by the study Genetics Committee):

Inheritance Pattern is Recessive and has at least 2 disease-causing variants which are homozygous or heterozygous in trans

OR

Inheritance Pattern is Recessive and has 2 disease-causing variants with unknown phase and meets all the following additional informatic criteria that is consistent with likely segregation in trans:

1. Investigator confirms genotype and phenotype are consistent with autosomal recessive inheritance
2. The 2 disease-causing variants have not been reported in cis in variant databases
3. No additional potentially pathogenic variants were found on the gene (and the sequencing data for the gene were sufficiently robust to detect any additional potentially pathogenic variants)
4. No potentially pathogenic variants were found in other common, likely candidate genes for the proposed condition

OR

Inheritance Pattern is Dominant, X-linked, or Mitochondrial and has at least 1 disease-causing variant

Both eyes must meet the following criteria at the Registry/Screening Visit to enroll into the genetic screening phase:

1. Both eyes must have a clinical diagnosis of retinal dystrophy
2. Both eyes must permit good quality photographic imaging (e.g., but not limited to, clear ocular media, adequate pupil dilation, stable fixation)

Exclusion Criteria:

Participants must not meet any of the following exclusion criteria at the Registry/Screening Visit to be eligible to enroll into the genetic screening phase:

1. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy including amiodarone, chloroquine, deferoxamine, hydroxychloroquine, pentosan polysulfate, tamoxifen, and deferoxamine Note: Since this is an observational study, pregnant women will not be specifically excluded from participation. However, minors that are pregnant shall be precluded from participation until they become the age of majority.

Ocular Exclusion Criteria:

If either eye has any of the following ocular exclusion criteria at the Registry/Screening Visit, then the participant is not eligible to enroll into the genetic screening phase:

1. Current vitreous hemorrhage
2. Current complications of pathological myopia (for example, but not limited to, myopic maculopathy including atrophy, scar, choroidal neovascularization, schisis) that could inhibit ability to obtain good quality photographic imaging
3. History of intraocular surgery (for example, but not limited to, cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within 3 months of Registry/Screening Visit
4. Current or any history of confirmed diagnosis of glaucoma (for example, but not limited to, glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery)
5. Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
6. History or current evidence of ocular disease that, in the opinion of the Investigator, may confound assessment of visual function (for example, but not limited to, tractional or rhegmatogenous retinal detachment, any vitreoretinal surgery, retinal vascular occlusion, proliferative diabetic retinopathy)
7. The following medications and treatments are prohibited as they can affect progression of retinitis pigmentosa (RP). The participant must not have received the following treatments:

   Any use of ocular stem cell or gene therapy Any treatment with ocriplasmin Treatment with Ozurdex (dexamethasone), Iluvien, or Yutiq (fluocinolone acetonide) intravitreal implant
8. The following medications and treatments are excluded within the specified timeframe:

Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Registry/Screening Visit date)

Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Registry/Screening Visit date is at least 5 times the half-life of the given product)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients with gene-related retinal degeneration. The universal registry is open to rare RD genes, to cross-sectionally characterize patients within rare RD genes (mild, moderate, and severe vision loss), so they are ready to be enrolled into a subsequent universal longitudinal natural history study as their gene is selected.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome: Characterize change using Visual field sensitivity measured with quantitative topographic analysis (hill of vision [HOV]) | Baseline and every year until study completion (4 years)
  Measured by Static Perimetry (SP) using Octopus 900 Pro
Functional Outcome: Characterize Change Using Early Treatment of Diabetic Retinopathy Study (ETDRS) / HOTV Best Corrected Visual Acuity (BCVA) letter score | Baseline and every year until study completion (4 years)
  Measured by Electronic Visual Acuity (EVA) system or ETDRS/HOTV charts
Functional Outcome: Characterize Change Using Low visual acuity test - for participants unable to see ETDRS letters | Baseline and every year until study completion (4 years)
  Measured by Berkeley Rudimentary Vision Test (BRVT) for Low Visual Acuity
Functional Outcome: Characterize Change Using ETDRS/HOTV best corrected low luminance visual acuity letter score | Baseline and every year until study completion (4 years)
  Measured by Electronic Visual Acuity (EVA) system or ETDRS/HOTV charts
Functional Outcome: Characterize Change in Mean retinal sensitivity | Baseline and every year until study completion (4 years)
  Measured by Fundus guided Microperimetry (MP) using MAIA
Functional Outcome: Characterize Change in Contrast sensitivity function | Baseline and every year until study completion (4 years)
  Measured by Contrast sensitivity CSV-1000E chart
Functional Outcome: Characterize Change in Retinal function using amplitudes and timing in response to rod- and cone-specific stimuli | Baseline and at study completion (4 years)
  Measured by Full-field Electroretinogram (ffERG) Diagnosys Espion
Functional Outcome: Characterize Change in Full-field retinal sensitivity | Baseline and every year until study completion (4 years)
  Measured by Full-field stimulus threshold (FST) testing to blue, white, and red stimuli using Diagnosys Espion
Functional Outcome: Characterize Change in Color vision function | Baseline and every year until study completion (4 years)
  Measured by Color vision testing using Lanthony D15
Structural Outcome: Characterize Change in Ellipsoid zone (EZ) area; outer nuclear layer and ganglion cell layer thicknesses | Baseline and every year until study completion (4 years)
  Measured by Spectral Domain Optical Coherence Tomography (SD-OCT) using Heidelberg Spectralis
Structural Outcome: Characterize Change Using Qualitative and quantitative assessments of autofluorescence pattern | Baseline and every year until study completion (4 years)
  Measured by Fundus Autofluorescence (FAF) using Optos

CONTACTS AND LOCATIONS:
Overall Officials: José-Alain Sahel, MD, Study Chair — Director, UPMC Eye Center University of Pittsburgh School of Medicine
Locations (36):
- United States (19):
  - University of Arkansas, Jones Eye Institute, Little Rock, Arkansas
  - USC Roski Eye Institute, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Emory Eye Center, Atlanta, Georgia
  - Johns Hopkins University, Wilmer Eye Institute, Baltimore, Maryland
  - Harvard Univ., Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Duke Eye Center, Durham, North Carolina
  - Oregon Health & Science Univ., Casey Eye Institute, Portland, Oregon
  - University of Pennsylvania, Scheie Eye Institute, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Alkek Eye Center, Houston, Texas
  - University of Utah, John Moran Eye Center, Salt Lake City, Utah
  - University of Wisconsin Madison, Madison, Wisconsin
  - Medical College of Wisconsin Eye Institute, Milwaukee, Wisconsin
- Centre for Eye Research Australia, East Melbourne, Victoria, Australia
- Ghent University, Ghent, Belgium
- Brazil (2):
  - INRET Clínica e Centro de Pesquisa, Belo Horizonte, Minas Gerais
  - Instituto de Genética Ocular, São Paulo, São Paulo Province
- Canada (3):
  - University of Alberta and Alberta Health Services, Edmonton, Alberta
  - University of Toronto, Hospital for Sick Children, Toronto, Ontario
  - University Health Network, Toronto
- Helsinki University Hospital, Helsinki, Finland
- CHNO des Quinze-Vingts, Paris, France
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- Vista Vision Eye Clinic, Brescia, Italy
- Retina and Genomics Institute, Yucatán, Merida, Mexico
- Radboud University Medical Center, Nijmegen, Netherlands
- Oslo University Hospital, Oslo, Norway
- Switzerland (2):
  - University Hospital Basel, Basel, Canton of Basel-City
  - University Hospital Jules-Gonin, Lausanne
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database is placed in the public domain on the FFB/Jaeb public website after the completion of each protocol and publication of the manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address

REFERENCES:
- See also: Foundation Fighting Blindness Public Website — https://public.jaeb.org/ffb
- See also: Uni-Rare Rare Gene List — https://s3.amazonaws.com/publicfiles.jaeb.org/UniRareGeneList2024.pdf

DOCUMENTS (1):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT05589714/Prot_002.pdf